CLINICAL TRIAL: NCT00787514
Title: Measurement of the Folate Receptor in Stored Plasma From Patients With Ovarian Cancer
Brief Title: FR in Stored Plasma
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Prof Stan Kaye, Institute of Cancer Research
Other Study IDs: CCR3029
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2008-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer, folate receptor, plasma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The folate receptor (FR) is a cell over expressed on the surface of certain cancers, this occurs most frequently in ovarian cancers. Some normal tissues also express the FR, however in these normal tissues, the FR is usually located on the tissue surface that is inaccessible to circulating drugs. As such, drugs which target the FR may potentially be used to target cancers which overexpress the FR while reducing toxicity to normal tissues. Therefore the ability to measure FR levels from different cancer types may help to select patients who are most likely to benefit from treatment with FR targeted therapies. Once such drug BGC945 is currently being tested in preclinical study at the Institute of Cancer Research

DETAILED DESCRIPTION:
FR may be released from the cancer cells in the blood. We have developed a method in the laboratory which has been able to measure the FR obtained from cancer cells in culture which has been added into blood. We would like to study if this method is able to measure the FR in stored plasma samples obtained from patients with ovarian cancer, so that it may be developed as a method for selecting patients for FR-target treatments such as BGC 945.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian cancer who have given informed consent to have blood collected for the plasma bank in the 'Pharmacogenetics and proteomics studies in patients receiving novel anticaner agents' study.

Exclusion Criteria:

* Patients who have withdrawn consent form their blood stored within the 'Pharmacogenetics and proteomics studies in patients receiving novel anticancer agents' study to be used for research.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the first stage of the study 13 samples will be analysed. If thee is one or more positive results the study will progress to the 2nd state to include 14 more samples.
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To measure the levels of soluble folate receptor in stored plasma obtained from patients with ovarian cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom